CLINICAL TRIAL: NCT03897881
Title: A Phase 2 Randomized Study of Adjuvant Immunotherapy With the Personalized Cancer Vaccine mRNA-4157 and Pembrolizumab Versus Pembrolizumab Alone After Complete Resection of High-Risk Melanoma (KEYNOTE- 942)
Brief Title: An Efficacy Study of Adjuvant Treatment With the Personalized Cancer Vaccine mRNA-4157 and Pembrolizumab in Participants With High-Risk Melanoma (KEYNOTE-942)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-4157-P201
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
Keywords: mRNA-4157; Individualized Neoantigen Therapy; INT; Pembrolizumab; Moderna
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-4157 and Pembrolizumab (Experimental): Participants will receive up to 9 doses of mRNA-4157 (every 21 days). Participants may continue on pembrolizumab (every 21 days) until disease recurrence, unacceptable toxicity, or they undergo up to 18 total cycles (approximately 1 year of treatment), whichever is sooner.
  Interventions: Drug: mRNA-4157; Biological: Pembrolizumab
- Pembrolizumab (Active Comparator): Participants will receive pembrolizumab (every 21 days) until disease recurrence, unacceptable toxicity, or they undergo up to 18 total cycles (approximately 1 year of treatment), whichever is sooner.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Drug: mRNA-4157 — Individualized Neoantigen Therapy
  Arms: mRNA-4157 and Pembrolizumab
Biological: Pembrolizumab — Intravenous infusion

SUMMARY:
The purpose of this study is to assess whether postoperative adjuvant therapy with mRNA-4157 and pembrolizumab improves recurrence free survival (RFS) compared to pembrolizumab alone in participants with complete resection of cutaneous melanoma and a high risk of recurrence.

ELIGIBILITY:
Key Inclusion Criteria:

* Resectable cutaneous melanoma metastatic to a lymph node and at high risk of recurrence
* Complete resection within 13 weeks prior to the first dose of pembrolizumab
* Disease free at study entry (after surgery) with no loco-regional relapse or distant metastasis and no clinical evidence of brain metastases
* Has an formalin fixed paraffin embedded (FFPE) tumor sample available suitable for sequencing
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Normal organ and marrow function reported at screening

Key Exclusion Criteria:

* Prior malignancy, unless no evidence of that disease for at least 5 years prior to study entry
* Prior systemic anti-cancer treatment (except surgery and interferon for thick primary melanomas. Radiotherapy after lymph node dissection is permitted)
* Live vaccine within 30 days prior to the first dose of pembrolizumab
* Transfusion of blood or administration of colony stimulating factors within 2 weeks of the screening blood sample
* Active autoimmune disease
* Immunodeficiency, systemic steroid therapy, or any other immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab
* Solid organ or allogeneic bone marrow transplant
* Pneumonitis or a history of (noninfectious) pneumonitis that required steroids
* Prior interstitial lung disease
* Clinically significant heart failure
* Known history of human immunodeficiency virus (HIV)
* Known active hepatitis B or C
* Active infection requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2032-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS), Assessed Using Radiological Imaging | Up to 7 years
  RFS is defined as the time between the date of first dose of pembrolizumab and the date of recurrence (local, regional, or distant metastasis), new primary melanoma, or death (whatever the cause), whichever occurs first.

SECONDARY OUTCOMES:
Distant Metastasis-Free Survival (DMFS), Assessed Using Radiological Imaging | Up to 7 years
  DMFS is defined as the time between the date of first dose of pembrolizumab and the date of the first distant metastasis or the date of death (whatever the cause), whichever occurs first.
Number of Participants With Adverse Events (AEs) | Baseline through 100 days after last mRNA-4157 dose or up to 90 days after the last dose of pembrolizumab, whichever is later (for mRNA-4157 and Pembrolizumab combination arm) and up to 90 days after last pembrolizumab dose (for Pembrolizumab only arm)
Number of Participants Who Discontinued Due to AEs | Baseline through 100 days after last mRNA-4157 dose or up to 90 days after the last dose of pembrolizumab, whichever is later (for mRNA-4157 and Pembrolizumab combination arm) and up to 90 days after last pembrolizumab dose (for Pembrolizumab only arm)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (17):
  - University of Arizona, Tucson, Arizona
  - California Pacific Medical Center Research Institute -CPMCRI, San Francisco, California
  - Angeles Clinic and Research Institute, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Smilow Cancer Center at Yale New Haven Hospital, New Haven, Connecticut
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - Northside Hospital, Atlanta, Georgia
  - UPMC Hillman Cancer Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Providence Cancer Institute, Portland, Oregon
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology PA, Dallas, Texas
- Australia (6):
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Affinity Clinical Research, Murdoch, Western Australia
  - One Clinical Research Perth, Murdoch, Western Australia
  - St John of God Hospital Subiaco, Subiaco, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weber JS, Carlino MS, Khattak A, Meniawy T, Ansstas G, Taylor MH, Kim KB, McKean M, Long GV, Sullivan RJ, Faries M, Tran TT, Cowey CL, Pecora A, Shaheen M, Segar J, Medina T, Atkinson V, Gibney GT, Luke JJ, Thomas S, Buchbinder EI, Healy JA, Huang M, Morrissey M, Feldman I, Sehgal V, Robert-Tissot C, Hou P, Zhu L, Brown M, Aanur P, Meehan RS, Zaks T. Individualised neoantigen therapy mRNA-4157 (V940) plus pembrolizumab versus pembrolizumab monotherapy in resected melanoma (KEYNOTE-942): a randomised, phase 2b study. Lancet. 2024 Feb 17;403(10427):632-644. doi: 10.1016/S0140-6736(23)02268-7. Epub 2024 Jan 18. PMID 38246194